CLINICAL TRIAL: NCT06496009
Title: The Clinical Characteristics and Efficacy of Immunotherapy in First-line PD-L1-negative Advanced NSCLC Patients: A Real-world Observational Study
Brief Title: The Clinical Characteristics and Efficacy of Immunotherapy in First-line PD-L1-negative Advanced NSCLC Patients
Acronym: LungCadX-RW
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2024LY0532
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: NSCLC
Keywords: NSCLC; PD-L1 negative; immunotherapy
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- immunotherapy group: advanced or metastatic non-small cell lung cancer who are PD-L1 negative and receiving first-line immunotherapy in routine clinical practice
  Interventions: Drug: PD-1 Inhibitors

INTERVENTIONS:
Drug: PD-1 Inhibitors — advanced or metastatic non-small cell lung cancer who are PD-L1 negative and receiving first-line immunotherapy in routine clinical practice
  Other Names: immunotherapy gourp

SUMMARY:
This study aims to include patients with advanced or metastatic non-small cell lung cancer who are PD-L1 negative and receiving first-line immunotherapy in routine clinical practice.

DETAILED DESCRIPTION:
This study aims to include patients with advanced or metastatic non-small cell lung cancer who are PD-L1 negative and receiving first-line immunotherapy in routine clinical practice. Clinical treatment of patients will not be intervened unless disease progression, intolerable toxicity, initiation of new anti-tumor therapy, withdrawal of informed consent, loss to follow-up, death, or other circumstances deemed appropriate by the investigator to discontinue treatment, whichever occurs first. The primary objective of the study is for investigators to assess the one-year progression-free survival (PFS) rate of immunotherapy as first-line treatment in PD-L1 negative advanced or metastatic NSCLC, evaluated according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before implementing any trial-related procedures;
* Aged 18-80 years;
* Wild-type EGFR/ALK;
* Patients with locally advanced (stage IIIb/IIIc), metastatic, or recurrent (stage IV) NSCLC confirmed by histology or cytology, who are not eligible for curative surgery and cannot undergo definitive radiotherapy/chemotherapy, according to the 8th edition of the TNM staging classification by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer;
* PD-L1 negative；
* Patients receiving first-line immunotherapy (such as PD-1/PD-L1 inhibitors).

Exclusion Criteria:

* The patient refused to join this study and declined follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced or metastatic non-small cell lung cancer who are PD-L1 negative and receiving first-line immunotherapy in routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 845 (Estimated)
Dates: Start 2024-07-08 (Estimated); Primary Completion 2026-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-Free Survival (PFS) rate | up to 12 month
  The 1-year Progression-Free Survival (PFS) rate is a clinical metric used to measure the percentage of patients who are still alive and have not experienced disease progression one year after the start of treatment.

SECONDARY OUTCOMES:
Progression-Free Survival | up to 24 months
  PFS is the length of time during and after treatment that a patient lives with the disease but it does not get worse. It is a standard measure used in clinical trials to evaluate the effectiveness of a treatment.
Overall Survival | up to 36 months
  OS refers to the length of time from either the date of diagnosis or the start of treatment that patients diagnosed with a disease are still alive
Objective Response Rate | up to 9 month
  Objective Response Rate (ORR) refers to the proportion of patients whose cancer shrinks (partial response) or disappears (complete response) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Su, PHD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
research article
Supporting Information: Study Protocol
Time Frame: up to 36 month
Access Criteria: Send an email requesting research